CLINICAL TRIAL: NCT04654455
Title: Prospective Study Evaluating Dry Eye in Patients Operated on for Ametropia by LASIK Surgery and Treated With REPADROP
Acronym: PREPADROP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1049
Record Dates: First submitted 2020-11-30; First posted 2020-12-04 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Describe the evolution of dry eye between 1 month and 3 months post-LASIK — Dry eye will be assessed through the OSDI (Ocular Surface Disease Index) questionnaire. The questionnaire will be dispensed during consultations by an orthoptist or an intern/junior doctor, at 1 month and at 3 months post-LASIK.

SUMMARY:
LASIK is a refractive surgery technique widely used in France. Postoperatively, the classic treatment after LASIK consists of instilling drops to reduce dry eyes. REPADROP® is an innovative eye drops stimulating corneal innervation. To date no study has quantified the improvement in dry eye syndrome and thus the quality of life of patients using REPADROP®.

ELIGIBILITY:
Inclusion Criteria:

Age over 18

* Planned bilateral LASIK surgery
* Use of Repadrop as postoperative eye drops
* Patient agreement to participate

Exclusion Criteria:

* History of corneal pathology
* Diabetes
* History of treatment with REPADROP® or CACICOL® or NGF® (other eye drops which are no longer available on the market to date but which would also improve corneal healing)
* Ongoing treatment with topical cyclosporine
* Presence of punctal plugs
* Adults who are the subject of a legal protection measure (guardianship, curators)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to hospital for LASIK surgery for ametropia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Variation in OSDI (Ocular Surface Disease Index) score | 3 Months
  Variation in OSDI (Ocular Surface Disease Index) score between 1 month and 3 months post-LASIK. The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, Rhone, France